CLINICAL TRIAL: NCT03231514
Title: Determining the Ergogenic Effects of Carb10™ Supplementation on Carbohydrate-Rich and Carbohydrate-Restricted Diets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Compound Solutions Inc. (Industry)
Responsible Party: Principal Investigator, Jordan Joy, Principal Investigator, Texas Woman's University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19151
Record Dates: First submitted 2017-07-12; First posted 2017-07-27 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Ketogenic Dieting
Keywords: body composition; exercise performance; keto-adaptation
MeSH Terms: interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Semi-randomized, parallel-group, single-blind diet and exercise intervention
Who Masked: Participant
Masking Description: Participants are blinded to the pre-workout drink content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Carbohydrate Diet & Placebo & Exercise (Placebo Comparator): This group receives the carbohydrate-based diet and flavored placebo pre-workout drink. All participate in the exercise intervention.
  Interventions: Other: Exercise
- Carbohydrate Diet & Carbohydrate Supplement(Carb10) & Exercise (Active Comparator): This group receives the carbohydrate-based diet and supplemental carbohydrate. Will be compared to Carbohydrate & Placebo for effects of supplement. All participate in the exercise intervention.
  Interventions: Dietary Supplement: Carbohydrate Supplement (Carb10); Other: Exercise
- Ketogenic Diet & Placebo & Exercise (Experimental): This group receives the ketogenic diet and flavored placebo. It is both an experimental (vs. carbohydrate diet & placebo) and placebo control group (vs. ketogenic & supplement). All participate in the exercise intervention.
  Interventions: Other: Diet; Other: Exercise
- Ketogenic Diet & Carbohydrate Supplement (Carb10) & Exercise (Experimental): This group receives the ketogenic diet and supplemental carbohydrate. All participate in the exercise intervention.
  Interventions: Dietary Supplement: Carbohydrate Supplement (Carb10); Other: Diet; Other: Exercise

INTERVENTIONS:
Dietary Supplement: Carbohydrate Supplement (Carb10) — 2 of 4 arms will be supplemented with carbohydrate pre-workout (Carb10, Compound Solutions, Carlsbad, CA)
  Arms: Carbohydrate Diet & Carbohydrate Supplement(Carb10) & Exercise; Ketogenic Diet & Carbohydrate Supplement (Carb10) & Exercise
Other: Diet — 2 groups will be on a carbohydrate-based diet (% energy from carbohydrate:fat:protein, 53:24:23) and 2 groups will be on a ketogenic diet (72:5:23)
  Arms: Ketogenic Diet & Carbohydrate Supplement (Carb10) & Exercise; Ketogenic Diet & Placebo & Exercise
Other: Exercise — All groups will participate in a standardized exercise intervention.

SUMMARY:
The study will examine the performance and body composition effects of ketogenic vs carbohydrate-based diets, determine the carbohydrate tolerance ("carbohydrate threshold") for active individuals on a ketogenic diet, and then, reexamine the performance and body composition effects when the diets are modified with supplemental carbohydrate up to the newly defined "ketogenic threshold."

DETAILED DESCRIPTION:
Participants will be recruited from TWU and the Denton area and grouped in a semi-randomized fashion that considers dietary preferences. They will then undergo baseline testing, begin the diet and training interventions, followed by post-testing (phase 1) and a carbohydrate titration period in the ketogenic diet group (phase 2). In the following academic semester, the training intervention will be repeated with an adjusted dietary carbohydrate level, delivered as a pre-workout supplement, corresponding to Phase 2 (Phase 3).

Phase 1 will consist of diets at an energy level estimated by the Mifflin St. Jeor equation adjusted by 1.625 for exercise. The exercise intervention will be a supervised, periodized (daily undulating), 9-week concurrent resistance (3 days/week) and cardiovascular (2 days/week) exercise program designed to improve body composition and performance variables. During phase 2, the ketogenic diet participants will continue exercising with the same program while consuming incrementally greater quantities of carbohydrate pre-workout until the state of ketosis is lost. Phase 3 will be identical to Phase 1, but diets will be modified to include more carbohydrate. As of completing Phase 2, this amount has been determined to be 20g of Carb10 (pea starch).

ELIGIBILITY:
Inclusion Criteria:

* consistently exercising at least 3 days per week for the past 2 years, participating in both cardiovascular and resistance exercise at least once per week for the past 2 years, reported themselves as healthy, and were willing and able to comply with study protocols

Exclusion Criteria:

* using tobacco of any form, a history of medical events, reporting any supplement or medication use that may affect study outcomes, regularly consuming > 7 alcoholic beverages per week, appearing unfit to handle the training program, inability to complete baseline testing, having a BMI > 35 kg/m2, or becoming < 80% compliant with training or dietary interventions.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Body Composition | 0 and 10 weeks
  Will be measured as fat and lean soft tissue mass in kg by dual x-ray absorptiometry (DXA)
Change in Anaerobic Cardiovascular Performance | 0 and 10 weeks
  Will be measured as peak and average power output in Watts during a repeated Wingate sprint test

SECONDARY OUTCOMES:
Change in Body Composition | 0 and 10 weeks
  In addition to DXA, body composition will be verified using bioelectric impedance (BIS) estimations of fat-free and fat mass in kg
Change in Body Water | 0 and 10 weeks
  BIS determined total, intra-, and extra-cellular fluid in Liters
Change in Cross-sectional Area | 0 and 10 weeks
  B-mode ultrasound determined cross-sectional area of the rectus femoris in cm squared
Change in Muscle Thickness | 0 and 10 weeks
  B-mode ultrasound determined combined thickness of the vastus lateralis and vastus medius in cm
Change in Aerobic Performance | 0 and 10 weeks
  measured as a 5km time trial with a 250m hill segment (8% grade) at 1km and 4km on a treadmill
Change in Vertical Jump Height | 0 and 10 weeks
  measured using vertec
Change in Vertical Jump Power | 0 and 10 weeks
  measured using linear force transducer
Change in Vertical Jump Velocity | 0 and 10 weeks
  measured using linear force transducer
Change in Vertical Jump Force | 0 and 10 weeks
  measured using linear force transducer
Change in Strength | 0 and 10 weeks
  measured as 1 repetition maximum
Change in Insulin | 0 and 10 weeks
  measured using clinical analyzer pmol/L
Change in HDL | 0 and 10 weeks
  measured using clinical analyzer mg/dL
Changes in LDL | 0 and 10 weeks
  measured using clinical analyzer mg/dL
Changes in Triglycerides | 0 and 10 weeks
  measured using clinical analyzer mg/dL
Changes in Aspartate Amino Transferase | 0 and 10 weeks
  measured using clinical analyzer U/L
Changes in Alanine amino Transferase | 0 and 10 weeks
  measured using clinical analyzer U/L
Changes in HbA1C | 0 and 10 weeks
  measured using clinical analyzer mmol/mol
Changes in Creatine Kinase | 0 and 10 weeks
  measured using clinical analyzer U/L
Changes in Total Testosterone | 0 and 10 weeks
  measured using ELISA ng/dL
Changes in Free Testosterone | 0 and 10 weeks
  measured using ELISA ng/dL
Changes in Total Estrogens | 0 and 10 weeks
  measured using ELISA pg/mL
Changes in Triiodothyronine | 0 and 10 weeks
  measured using ELISA ng/dL
Changes in Thyroxine | 0 and 10 weeks
  measured using ELISA ng/dL
Changes in Thyroid Stimulating Hormone | 0 and 10 weeks
  measured using ELISA mu/L
changes in C-reactive Protein | 0 and 10 weeks
  measured using ELISA mg/L
Changes in Dehydroepiandrosterone sulfate | 0 and 10 weeks
  measured using ELISA ug/dL
Changes in Sex hormone Binding Globulin | 0 and 10 weeks
  measured using ELISA nmol/L
Changes in Cortisol | 0 and 10 weeks
  measured using ELISA ug/dL
Changes in Whole Blood Betahydroxybutyrate | about every 3-7 days
  measured using handheld meter mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Joy, MS, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Volek JS, Freidenreich DJ, Saenz C, Kunces LJ, Creighton BC, Bartley JM, Davitt PM, Munoz CX, Anderson JM, Maresh CM, Lee EC, Schuenke MD, Aerni G, Kraemer WJ, Phinney SD. Metabolic characteristics of keto-adapted ultra-endurance runners. Metabolism. 2016 Mar;65(3):100-10. doi: 10.1016/j.metabol.2015.10.028. Epub 2015 Nov 2. PMID 26892521
- [Background] Wilson JM, Lowery RP, Roberts MD, Sharp MH, Joy JM, Shields KA, Partl JM, Volek JS, D'Agostino DP. Effects of Ketogenic Dieting on Body Composition, Strength, Power, and Hormonal Profiles in Resistance Training Men. J Strength Cond Res. 2020 Dec;34(12):3463-3474. doi: 10.1519/JSC.0000000000001935. PMID 28399015
- [Background] Burke LM, Ross ML, Garvican-Lewis LA, Welvaert M, Heikura IA, Forbes SG, Mirtschin JG, Cato LE, Strobel N, Sharma AP, Hawley JA. Low carbohydrate, high fat diet impairs exercise economy and negates the performance benefit from intensified training in elite race walkers. J Physiol. 2017 May 1;595(9):2785-2807. doi: 10.1113/JP273230. Epub 2017 Feb 14. PMID 28012184
- [Background] Urbain P, Strom L, Morawski L, Wehrle A, Deibert P, Bertz H. Impact of a 6-week non-energy-restricted ketogenic diet on physical fitness, body composition and biochemical parameters in healthy adults. Nutr Metab (Lond). 2017 Feb 20;14:17. doi: 10.1186/s12986-017-0175-5. eCollection 2017. PMID 28239404